CLINICAL TRIAL: NCT05531708
Title: Safety and Efficacy Study of Novel Mesothelin CAR-T Cell Therapy in Patients With Mesothelin-positive Advanced Refractory Solid Tumors
Brief Title: Exploratory Study of Novel MSLN CAR-T Cell Therapy in Patients With MSLN-positive Advanced Refractory Solid Tumors
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: The study is not initiated and we want it to be withdrawn.
Sponsor: Shanghai Pudong Hospital (Other)
Collaborators: UTC Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-IIT-004-E02
Record Dates: First submitted 2022-08-22; First posted 2022-09-08 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Mesothelin-positive Advanced Refractory Solid Tumors
Keywords: Anti-mesothelin CAR-T; Solid tumor
MeSH Terms: interventions — fludarabine; fludarabine phosphate; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anti-mesothelin CAR-T cells (Experimental): A conditioning chemotherapy regimen of fludarabine and cyclophosphamide will be administered followed by investigational treatment, anti-mesothelin CAR-T cells.
  Interventions: Biological: Anti-mesothelin CAR-T cells; Drug: Fludarabine; Drug: Cyclophosphamide

INTERVENTIONS:
Biological: Anti-mesothelin CAR-T cells — D0: Anti-mesothelin CAR-T cells are autologous genetically modified T cells. Cells will be infused intravenously.
Drug: Fludarabine — D-7 to D-3: Fludarabine (25 mg/m^2/day) will be administered intravenously for 5 days.
  Other Names: Fludara
Drug: Cyclophosphamide — D-7 and D-6: Cyclophosphamide (60 mg/kg/day) will be administered intravenously for 2 days.
  Other Names: Cytoxan

SUMMARY:
This is a single-arm, open-label, exploratory clinical study to evaluate the safety and efficacy of novel Mesothelin CAR-T in patients with Mesothelin-positive advanced refractory solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Solid tumors positive for the Mesothelin antigen by Immunohistochemistry/Immunocytochemistry (IHC/ICC); histological diagnosis of malignancy refractory to, or relapsing after standard therapy.
2. At least one measurable lesion according to RECIST v1.1.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
4. Life expectancy ≥ 3 months.
5. Neutrophils ≥ 1.0×10^9/L; Lymphocytes ≥ 0.5×10^9/L; Hemoglobin ≥ 80 g/L; Platelets ≥ 75×10^9/L.
6. Adequate hepatic, renal, cardiac and coagulation function defined as:

   * Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) ≤ 2.5 × upper limit of normal (ULN); patients with liver metastasis must be ≤ 5 × ULN;
   * Total bilirubin (TBIL) ≤ 1.5 × ULN; TBIL of patients with Gilbert's Syndrome must less than 3.0 mg/dL;
   * Serum creatinine (Cr) ≤ 1.5 × ULN, and creatinine clearance rate (Ccr) ≥ 60 mL/min;
   * Left ventricular ejection fraction (LVEF) > 45%;
   * Prothrombin time (PT) and activated partial thromboplastin time (APTT) ≤ 1.5 × ULN.
7. Negative screen for infectious disease markers including HIV-Ab, HCV-Ab, HBeAg, HBsAg, and syphilis. Note - Participants with history of prior HBV infection are eligible if the HBV viral load is undetectable. Participants with a history of HCV infection who were treated for hepatitis C and cured are eligible if hepatitis C viral load is undetectable.
8. The toxicities from any prior therapy must have recovered to a grade 1 or less (except for toxicities such as alopecia or vitiligo) according to NCI CTCAE v5.0.
9. The washout period of previous treatment:

   * Cytotoxic chemicals, monoclonal antibodies or immunotherapy should be washed out for at least 4 weeks before leukapheresis; anti-CTLA-4 antibodies should be washed out for at least 6 weeks;
   * Systemic corticosteroids or other immunosuppressive therapies should be washed out for at least 2 weeks before leukapheresis;
   * Biologicals or other approved molecular targeted inhibitors should be eluted for at least 1 week or 5 half-lives (whichever is longer) prior to leukapheresis.
10. Participants must be able to understand the protocol and be willing to enroll the study, sign the informed consent, and be able to comply with the study and follow-up procedures.

Exclusion Criteria:

1. Patients with central nervous system involvement.
2. Patients with clinically significant systemic disease (such as: severe active infection or significant cardiac, pulmonary, hepatic, nervous system, or other organ dysfunction) that evaluated by the investigator would impair the patient's ability to tolerate the treatments used in this study or significantly increase the risk of complications.
3. Any known or suspected autoimmune disease; or active, chronic or recurrent immune-mediated disease (within one year prior to enrollment) requiring steroid or other immunosuppressive therapy.
4. History of severe systemic hypersensitivity reaction to the drugs/ingredients used in this study.
5. Have received any allogeneic tissue/organ transplantation (including bone marrow transplantation, stem cell transplantation, liver transplantation, kidney transplantation), except for the transplantation that does not require immunosuppressive therapy (such as: corneal transplantation, hair transplantation.)
6. Have received any genetic engineering modified T cell therapy (including CAR-T, TCR-T).
7. History of major surgery and unrecovered severe trauma within 4 weeks prior to signing informed consent.
8. History of another malignancy tumor, except for non-melanoma skin cancer and carcinoma in situ of bladder, stomach, colon, cervix/dysplasia, melanoma, or breast.
9. History of neuropsychiatric diseases diagnosed by the ICD-11 criteria or evaluated by investigator.
10. For any other reasons, the patients are believed not suitable for participation in this study by investigators.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-04-02 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
TEAEs | 4 weeks after the CAR-T cells infusion
  Incidence and severity of treatment emergent adverse events.
TRAEs | 4 weeks after the CAR-T cells infusion
  Incidence and severity of treatment related adverse events.
AESIs | 4 weeks after the CAR-T cells infusion
  Incidence and severity of AEs of special interest.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) (PR+CR) | 12 weeks
  The proportion of participants with complete response(CR) or partial response(PR) as measured by RECIST 1.1 criteria.
Duration of Overall Response（DOR） | 24 months
  Time from documentation of disease response to disease progression.

CONTACTS AND LOCATIONS:
Overall Officials: Zhiguo Long, Principal Investigator — Shanghai Pudong Hospital
Locations (1):
- Shanghai Pudong Hospital, Fudan University Affiliated Pudong Medical Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No